CLINICAL TRIAL: NCT06533358
Title: An Open-label, Sequential Dose Escalation/De-escalation Clinical Trial of MT1002 in Subjects With Acute Coronary Syndrome Undergoing PCI
Brief Title: A Clinical Study of MT1002 in Subjects With Acute Coronary Syndrome Undergoing PCI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shaanxi Micot Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT1002-II-C04
Record Dates: First submitted 2024-07-18; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MT1002 Injection (Experimental): MT1002 is infused once only, once for 4h
  Interventions: Drug: MT1002 Injection

INTERVENTIONS:
Drug: MT1002 Injection — MT1002 is infused once only, once for 4h. MT1002 is for subjects with acute coronary syndrome undergoing PCI
  Other Names: No other name

SUMMARY:
An Open-label, Sequential Dose Escalation/De-escalation Clinical Trial of MT1002 in Subjects With Acute Coronary Syndrome Undergoing PCI.

DETAILED DESCRIPTION:
MT1002 is a novel 32-amino acid synthetic peptide aimed to combine molecular functions of both a direct thrombin inhibitor and a platelet glycoprotein IIb/IIIa receptor antagonist, indicated for use as an antithrombotic and anticoagulant in patients with ACS and in patients undergoing PCI.

This study is an Open-label, sequential dose escalation/de-escalation clinical trial of MT1002 in subjects with acute coronary syndrome undergoing PCI. First dose cohort is 0.60 mg/kg (initial loading dose, intravenous bolus) + 1.2 mg/kg/h*4 h (maintenance dose, intravenous infusion). The Safety Review Committee makes decisions on subsequent dose adjustments. Dose escalation/de-escalation and stopping rules have been put in place to ensure the safety of the patients in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female aged 18-85 years old (both 18 and 85 years old)
2. Diagnosis of acute coronary syndrome (ACS)
3. Subjects who will undergo PCI during hospitalization
4. Able to understand and willing to sign written informed consent prior to undertaking any study-related activities
5. Females of childbearing potential must have a negative pregnancy test result prior to enrollment or be postmenopausal for at least 1 year, or permanently sterilized for ≥ 6 weeks. For women of childbearing potential and men with female partners of childbearing potential, effective contraception must be used if they are sexually active from the time of informed consent until 90 days after MT1002 administration

Exclusion Criteria:

1. cardiogenic shock, or cardiopulmonary resuscitation (CPR）
2. Suspicious aortic dissection, pericarditis, endocarditis
3. Has any history of intracranial hemorrhage or structural abnormalities
4. Transient ischemic attack, stroke within 6 months
5. History of gastrointestinal or genitourinary bleeding within 1 month
6. Major surgery within 1 month
7. The following surgeries are planned within 1 month of enrollment: CABG, valve surgery, or other invasive procedures
8. Long-term treatment with non-steroidal anti-inflammatory drugs (except aspirin), cyclooxygenase (COX)-2 inhibitors, within 1 month prior to screening
9. Prior (within 7 days prior to enrollment) or planned use of thrombolytic agents, bivalirudin, or fondaparinux. 12 hours before enrollment, unfractionated heparin or low molecular weight heparin was injected subcutaneously.
10. Use of coumarin derivatives and/or factor Xa inhibitors in the past 7 days
11. Anticipated need for oral anticoagulants within 3 days of dosing
12. Severe uncontrolled hypertension persists even within 24 hours of adequate treatment
13. According to the judgment of the investigator, the subject has a high risk of bleeding, such as active bleeding, bleeding tendency, coagulation disorders, etc
14. Known associated hematologic abnormalities
15. Known to have a malignancy or comorbid other disease that may lead to protocol non-adherence with a life expectancy of < 1 year
16. Known severe liver disease
17. Known hepatitis B and hepatitis C, HIV screening serology positive, except for the low viral replication phase.
18. Known chronic kidney disease
19. Known allergy or intolerance to aspirin, clopidogrel, ticagrelor, prasugrel, bivalirudin, unfractionated heparin, P2Y12 antagonists, or contrast agents.
20. Weight: male subjects should not be less than 50.0kg, female subjects should not be less than 45.0kg, and body mass index within the range of 18.0~30.0kg/m2 (including boundary values)
21. Subjects who have previously used MT1002.
22. Unable to fully cooperate with the study protocol.
23. Has any other medical or psychiatric illness that, in the opinion of the investigator, precludes participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
percentage of subjects who achieved target ACT (200-300 s) | Day 1, 24 hours （Day 2） to Day 30±2 after intravenous injection on Day 1
  percentage of subjects achieving target ACT (200-300 s) among subjects receiving MT1002 (not switching to standard care) pre/intraoperatively and after successful PCI
Major bleeding events | Day 1 to end of follow-up period (Day 30±2)
  Adverse events (AEs): Major bleeding events (Bleeding Academic Research Consortium [BARC] type 3-5)

CONTACTS AND LOCATIONS:
Overall Officials: Changsheng Ma, Medical phd, Principal Investigator — Beijing Anzhen Hospital Affiliated to Capital Medical University
Locations (2):
- China (2):
  - Beijing Anzhen Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Xianyang Hospital, Yan'an University, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: No